CLINICAL TRIAL: NCT06550323
Title: Göğüs Tüpü Çıkarma İşlemi Sırasında Sanal Gerçeklik Uygulamasının Ağrı, Anksiyete ve Konfora Etkisi
Brief Title: Effect of Virtual Reality Application on Pain, Anxiety and Comfort During Chest Tube Removal Procedure
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hale Rumeysa Seçer (Other)
Responsible Party: Sponsor-Investigator, Hale Rumeysa Seçer, Nurse, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: VRA15
Record Dates: First submitted 2024-07-20; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Chest Tube Removal
Keywords: virtual reality; pain; anxiety; comfort
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group using virtual reality glasses (Experimental): Virtual reality application will be applied to this group and virtual reality glasses will be put on 5 minutes before the procedure and the video will be started to be watched during the process.
  Interventions: Device: Group using virtual reality glasses
- Group not using virtual reality glasses (No Intervention): Standard protocols will be applied to this group and no action will be taken.

INTERVENTIONS:
Device: Group using virtual reality glasses — Group using virtual reality glasses: During the procedure, individuals will wear glasses.
  Arms: Group using virtual reality glasses

SUMMARY:
Chest tubes are used to eliminate possible acute or chronic problems that may occur after trauma or surgical interventions to the chest area. This process, which aims to drain the fluid, blood or air accumulated in the pleural area, works with the support of closed underwater drainage systems. The chest tubes, which remain in place for a long time, fuse with the endothelium lying in the chest cavity. For this reason, the adhesions formed with the fusion cause very severe acute pain in the patient with the pulling force applied during removal.The high level of pain of the person will cause an increase in the level of anxiety and a decrease in the level of comfort. The anxiety experienced by the patients will also reduce the tolerance to pain.It has been observed that the use of virtual reality in the field of health significantly reduces the level of pain and anxiety during medical procedures, shortens wound healing and hospital stay, and increases compliance with treatment.In the literature, no studies were found in which the effects of virtual reality application on pain, anxiety and comfort were evaluated in patients whose chest tube was removed.Thereforee, this study was conducted to evaluate the effect of virtual reality application against all these negative situations.

ELIGIBILITY:
* Study Inclusion Criteria:

  * Must be between the ages of 18-65,
  * Must have undergone coronary artery bypass graft surgery and have a chest tube,
  * Must participate in the study voluntarily,
  * Must not have vision or hearing problems,
  * Must not have disorientation in place and time,
  * Must not have any psychiatric disorders,
* Study Exclusion Criteria:

  * Those with chronic pain and routinely using painkillers,
  * Those using painkillers before the procedure,
  * Those with problems such as migraine, vertigo, dizziness,
  * Patients using prescription glasses and those having vision problems without glasses were not included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
visual analog scale | 5 month
  To evaluate pain severity, pain results are evaluated by scoring between 0-10. While 0 indicates "No pain", 10 indicates "Unbearable pain".
  The minimum value is 0 and the maximum value is 10. 0 represents a good result and 10 represents a bad result
State-Trait Anxiety Inventory Scale | 5 month
  It is a 4-point Likert-type scale with 40 items and is scored as "never": 1, "a little": 2, "a lot": 3, "completely": 4, according to the degree of severity of the feelings, thoughts or behaviors expressed by the items. anxiety level will be determined.
comfort scale | 5 month
  It is a scale ranging from 0 to 10 points. While 0 points indicate 'most comfortable', 10 points indicate 'most uncomfortable'.
  The minimum value is 0 and the maximum value is 10. 0 represents a good result and 10 represents a bad result
verbal pain scale | 5 month
  0 points indicate "No pain", 1 point indicates "Mild pain", 2 points indicate "Moderate pain" and 3 points indicate "Severe pain".

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Derived] Secer H, Yayla A. The effects of virtual reality on pain, anxiety, and comfort during the chest tube removal procedure: A randomized clinical trial. Complement Ther Clin Pract. 2025 Feb;58:101931. doi: 10.1016/j.ctcp.2024.101931. Epub 2024 Nov 8. PMID 39541838